CLINICAL TRIAL: NCT05580796
Title: Investigator Initiated Clinical Trial on the Tolerance, Safety and Preliminary Efficacy of KSH01-TCRT Injection in Solid Tumor Subjects
Brief Title: KSH01-R02-101 Solid Tumors
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: TCRx Therapeutics Co.Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KSH01-R02-101
Record Dates: First submitted 2022-10-08; First posted 2022-10-14 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Solid Tumor
Keywords: Genetic engineering of T-cells

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TCR-T cells (Experimental): TCR-T cell injection
  Interventions: Drug: KSH01 injection

INTERVENTIONS:
Drug: KSH01 injection — TCR-T cell injection

SUMMARY:
1. . safety and tolerance
2. . objective response rate

DETAILED DESCRIPTION:
1. . To evaluate the safety and tolerance of autologous TCR-T cells in target positive solid tumor patients.
2. . Preliminary evaluation of objective response rate (ORR) of autologous TCR-T cells in target positive solid tumor patients (such as esophageal cancer, gastric cancer, head and neck cancer, bladder cancer, melanoma, sarcoma, etc.)

ELIGIBILITY:
Inclusion Criteria:

* 1) Voluntary participation in clinical research; Fully understand the study and voluntarily sign the informed consent form; Willing to follow and able to complete all test procedures;
* 2) Male or female, 18 to 70 years old (including boundary value);
* 3) Malignant solid tumors failed to receive standard treatment;
* 4) HLA-A * 02 is positive and tumor target is positive (the staining intensity of target tumor cells is divided into 0, 1+, 2+, 3+, and more than 30% of cancer cells express 2+or 3+positive as the target is positive)
* 5). All toxic reactions caused by previous anti-tumor treatment are alleviated to grade 0-1 (according to NCI CTCAE version 5.0) or to an acceptable level of inclusion/exclusion criteria. Other poisons such as alopecia and vitiligo that researchers believe do not pose a safety risk to subjects
* 6) There is sufficient organ function (no medical support such as blood transfusion and granulocyte colony stimulating factor within 14 days before cell transfusion), which is defined as follows:
* 6.1) Blood system:
* 6.1.1) Neutrophil count (ANC) is not lower than the lower limit of normal value of the center;
* 6.1.2) White blood cell (WBC) shall not be lower than the lower limit of normal value of the center;
* 6.1.3) Platelet count (PLT) shall not be lower than the lower limit of normal value of the center;
* 6.1.4) Hemoglobin (Hb) shall not be lower than 0.8 * LLN (lower limit of normal value);
* 6.2) Liver function:
* 6.2.1) Total bilirubin (TBIL) ≤ 2.0 × Upper limit of normal (ULN), Gilbert disease subjects should be ≤ 3 × ULN；
* 6.2.2) AST, ALT ≤ 3 × ULN (in the dose expansion stage, the subjects with liver metastasis or liver cancer can be ≤ 5 × ULN）； Alkaline phosphatase (ALP) ≤ 2.5 × ULN (bone metastasis subject, ALP ≤ 5 × ULN）；
* 6.3) Renal function:
* 6.3.1) Serum creatinine ≤ 1.5 × ULN or creatinine clearance ≥ 50 ml/min (Cockcroft Gault formula: ([140 age] × Weight [kg] × [0.85 for women only])/(72 × Creatinine (mg/dl));
* 6.3.2) Qualitative urine protein ≤ 1+; If the urine protein is qualitative ≥ 2+, a 24-hour urine protein quantitative test is required. If the 24-hour urine protein quantitative test is less than 1 g, it is acceptable;
* 6.4) Coagulation function: those not receiving anticoagulation treatment: International normalized ratio (INR), activated partial thromboplastin time (APTT) should be ≤ 1.5 × ULN； Subjects with liver metastasis or liver cancer should be ≤ 2 × ULN；
* 7) Physical condition: The score of the Eastern American Cooperative Oncology Group (ECOG) was 0-1;
* 8) Expected survival time ≥ 12 weeks;
* 9) According to RECIST 1.1, there is at least one measurable lesion (dose expansion stage) or evaluable lesion (dose increase stage);
* 10) After evaluation, enough PBMC cells can be collected from the subjects to prepare autologous TCR-T cells;
* 11) After evaluation, the prepared autologous TCR-T cells are sufficient in quantity and qualified in quality, and can be used for clinical reinfusion of corresponding dose;
* 12) The blood pregnancy result of female subjects with fertility within 3 days before cell transfusion was negative, and they were willing to sign informed consent from the end of the last medication to 6 months, keep abstinence or take medically approved effective contraceptive measures (such as intrauterine device, pregnancy avoidance device);
* 13) Male subjects are willing to keep abstinence or take medically approved effective contraceptive measures within 6 months from signing the informed consent form to the end of the last medication, and do not donate sperm during this period;
* 14) All subjects should provide tumor tissue samples that can be used for target analysis, which should be archived samples or fresh biopsy samples (bone biopsy samples are not accepted). Only those with positive target expression can enter the study.

Exclusion Criteria:

* 1) History of serious allergic diseases, allergic history of serious drugs (including non marketed test drugs) or known allergy to any component of the proposed drugs (including pre-treatment drugs) in this protocol;
* 2) Previous coronary artery reconstruction;
* 3) Evidence of major haemorrhagic disorder or other obvious bleeding risks:
* 3.1) Previous history of intracranial hemorrhage or intracerebral hemorrhage;
* 3.2) The tumor focus invades large vessels and has obvious risk of bleeding;
* 3.3) Thrombosis or embolism occurred within 6 months before cell transfusion;
* 3.4) Clinically significant hemoptysis or tumor hemorrhage occurred within 1 month before cell transfusion;
* 3.5) Anticoagulant therapy (except low molecular weight heparin) for therapeutic purposes was used within 2 weeks before cell transfusion;
* 3.6) Within 10 days before cell reinfusion, they have used antiplatelet drugs, such as aspirin (>325 mg/day), clopidogrel (>75 mg/day), dipyridamole, ticlopidine or cilostazol;
* 4) Have received the following treatments or drugs before cell reinfusion:
* 4.1) Unhealed wound, ulcer or fracture within 28 days before cell reinfusion;
* 4.2) Inoculate live attenuated vaccine within 28 days before cell reinfusion;
* 4.3) The cells were treated with nitrosourea or mitomycin C within 6 weeks before reinfusion; Oral fluorouracil therapy was received 2 weeks before cell reinfusion or within 5 half lives of the drug (whichever is longer);
* 4.4) Within 2 weeks before cell reinfusion, the patient has received corticosteroids, or it is estimated that corticosteroids may be required during blood collection, cell collection or cell reinfusion; Except for the following cases: short-term (≤ 7 days) prednisone with a dose not higher than 10 mg/d or equivalent dose is used to prevent or treat non autoimmune conditions; Corticosteroids for local, nasal, intraocular, articular cavity or inhalation;
* 5) It is known that there is leptomeningeal metastasis, or uncontrolled or symptomatic central nervous system metastasis, with clinical symptoms, brain edema, spinal cord compression and/or progressive growth. Subjects with a history of central nervous system metastasis or spinal cord compression can be accepted if they have definitely received treatment and stopped using anticonvulsants and steroids 8 weeks before cell reinfusion, and their clinical manifestations are determined to be stable by the investigator;
* 6) Presence of any form of primary immunodeficiency;
* 7) Presence of any active autoimmune disease, Or asthmatic subjects who have a history of autoimmune diseases and are expected to relapse (including but not limited to: systemic lupus erythematosus, rheumatoid arthritis, psoriasis, multiple sclerosis, inflammatory bowel disease, and asthma requiring medical intervention with bronchodilators. The following cases are excluded: type 1 diabetes; skin diseases that do not require systemic treatment [such as vitiligo, psoriasis, alopecia] ； Hypothyroidism requiring only hormone replacement therapy; Asthma that has been completely relieved in childhood does not need any intervention in adulthood; Or other patients who are expected to have no relapse under the condition of no external trigger);
* 8) Within 6 months before cell reinfusion, the following conditions occurred: myocardial infarction, severe/unstable angina, arrhythmia with clinical significance and requiring clinical intervention, cerebrovascular accident/stroke, transient ischemic attack, subarachnoid hemorrhage, and cardiac insufficiency with NYHA grade ≥ II;
* 9) At present, there are uncontrollable pleural, pericardial and peritoneal effusion;
* 10) Before cell reinfusion, there were:
* 10.1) congenital long QT syndrome
* 10.2) pacemaker use
* 10.3) left ventricular ejection fraction (LVEF)<50%
* 10.4) QTcF interval>480 msec (QTcF=QT/(RR ^ 0.33)
* 10.5) cardiac troponin I or T>2.0 ULN
* 10.6) poorly controlled diabetes mellitus (fasting glucose ≥ 13.3 mM)
* 10.7) poorly controlled hypertension (systolic pressure ≥ 160 mmHg and/or diastolic pressure ≥ 100 mmHg);
* 10.8) Forced expiratory volume in the first second (FEV1) ≤ 60% or oxygen therapy is required;
* 11) During screening or before cell reinfusion, fever of unknown cause occurred>38.5 ° C (according to the judgment of the investigator, fever caused by tumor can be included in the group);
* 12) History of allograft transplantation is known;
* 13) Known history of alcohol abuse, psychotropic substance abuse or drug abuse;
* 14) Have a clear history of neurological or mental disorders, such as epilepsy, dementia, schizophrenia, etc;
* 15) Known to have acquired immunodeficiency syndrome (AIDS);
* 16) Serious active virus, bacterial infection or uncontrolled systemic fungal infection are known;
* 17) Virology test results (HIV, CMV, HSV, HPV, EBV, syphilis) are positive;
* 18) HBsAg positive or HBcAb positive, and HBV-DNA>200 IU/mL; HCV Ab is positive, and HCV RNA is higher than the lower detection limit of the research center;
* 19) According to the judgment of the investigator, the basic condition of the subject may increase the risk of receiving the test drug treatment, or the interpretation of the toxic reaction and adverse event may cause confusion;
* 20) It is expected to receive any other form of anti-tumor drug treatment during the study period;
* 21) Women in pregnancy or lactation;
* 22) Other investigators consider it inappropriate to participate in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-10-11 (Actual); Primary Completion 2025-10-11 (Estimated); Study Completion 2027-10-11 (Estimated)

PRIMARY OUTCOMES:
Number of participants in treatment related adverse events assessed by CTCAE v4.0 | about 3 years
  To evaluate the safety and tolerance of autologous TCR-T cells in target positive solid tumor subjects.
objective remission rate | about 3 years
  To preliminarily evaluate the objective remission rate of autologous TCR-T cells in the treatment of target positive solid tumor subjects (such as esophageal cancer, gastric cancer, head and neck cancer, bladder cancer, melanoma, sarcoma, etc.).

SECONDARY OUTCOMES:
Maximum tolerable dose values | about 3 years
  Maximum tolerable dose values
Changes in tumor size and time. | about 5 years
  Preliminary evaluation of anti-tumor efficacy of autologous TCR-T cells in solid tumor subjects
Concentration of pharmacokinetic values in plasma | about 3 years
  To evaluate the pharmacokinetics of autologous TCR-T cells in solid tumor subjects
Concentration of cytokine level value in plasma | about 3 years
  To evaluate the cytokine level of autologous TCR-T cells in solid tumor patients during treatment
Concentration of biomarker value in plasma | about 3 years
  Evaluation of biomarker characteristics of autologous TCR-T cells in solid tumor subjects

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese People's Liberation Army (PLA) General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No